CLINICAL TRIAL: NCT05840926
Title: Possible Prophylactic Role of the S. Salivarius K12 Probiotic Strain for the Upper Respiratory Tract Infection and Nursery-age Children
Brief Title: Probiotic S. Salivarius K12 for the Prevention of Upper Respiratory Tract Infection in Nursery-age Children
Acronym: PUNK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor, Liaquat University of Medical & Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LUMHS/REC/181
Record Dates: First submitted 2023-04-01; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Streptococcus salivarius K12 Treatment Group (Experimental): Children treated with Probiotic Streptococcus salivarius K12 Treatment for continuous 3-months
  Interventions: Dietary Supplement: Probiotic Streptococcus salivarius K12
- Control Group (Active Comparator): Children who did not receive any probiotic treatment
  Interventions: Other: No probiotic supplementation

INTERVENTIONS:
Dietary Supplement: Probiotic Streptococcus salivarius K12 — Oral 1 billion CFU of Probiotic Streptococcus salivarius K12
  Arms: Probiotic Streptococcus salivarius K12 Treatment Group
Other: No probiotic supplementation — Children who did not receive any probiotic supplementation
  Arms: Control Group

SUMMARY:
The purpose of this retrospective study is to assess the treatment benefits of probiotic Streptococcus salivarius K12 for the prevention of recurrent bacterial and viral infections of the pharynx, tonsils and ears in children under 3 years of age.

DETAILED DESCRIPTION:
Recurrent bacterial and viral infections of the pharynx, tonsils and ears are a problem that can affect children of all ages. The persistence of these infections can lead to an overuse of drugs such as antibiotics, antipyretics and anti-inflammatories, with the possible consequent presence of side effects and above all an increase in antibiotic resistance, a global public health issue.

In search at reducing the use of antibiotics and antivirals, there is currently a great scientific interest in probiotic therapies for the oral cavity infection.

The aim of this retrospective, controlled, multicenter, non-profit study is to evaluate the efficacy and safety of the administration of Streptococcus salivarius K12 in pediatric patients attending the 1st or 2nd year of nursery school (< 3 years of age ), in the prophylaxis of the most common bacterial or viral respiratory infections, assessing the consequent reduction in the use of antibiotics, antivirals or other therapies compared to children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children attending the 1st or 2nd year of nursery (under aged 3 years)
* Treated with probiotic Streptococcus salivarius K12 (1 billion CFU) for 90 continuous days
* Children not treated with probiotic Streptococcus salivarius K12

Exclusion Criteria:

* Children with underlying health condition

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 287 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of any Gastrointestinal upset | 03 Months
  Safety and tolerability of the probiotic treatment
Bacterial or respiratory viral infection | 03 Months
  Evaluation of the frequency of bacterial or respiratory viral infection
Use of antibiotics or antivirals | 03 Months
  Evaluation of the frequency of use of antibiotic or antiviral therapies

SECONDARY OUTCOMES:
Other pathologies | 03 Months
  Evaluation of the frequency of incidence of other pathologies such as GI

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University Hospital, Jāmshoro, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Pierro F, Risso P, Poggi E, Timitilli A, Bolloli S, Bruno M, Caneva E, Campus R, Giannattasio A. Use of Streptococcus salivarius K12 to reduce the incidence of pharyngo-tonsillitis and acute otitis media in children: a retrospective analysis in not-recurrent pediatric subjects. Minerva Pediatr. 2018 Jun;70(3):240-245. doi: 10.23736/S0026-4946.18.05182-4. Epub 2018 Jan 11. PMID 29322750
- [Background] Sarlin S, Tejesvi MV, Turunen J, Vanni P, Pokka T, Renko M, Tapiainen T. Impact of Streptococcus salivarius K12 on Nasopharyngeal and Saliva Microbiome: A Randomized Controlled Trial. Pediatr Infect Dis J. 2021 May 1;40(5):394-402. doi: 10.1097/INF.0000000000003016. PMID 33298762
- [Background] Burton JP, Cowley S, Simon RR, McKinney J, Wescombe PA, Tagg JR. Evaluation of safety and human tolerance of the oral probiotic Streptococcus salivarius K12: a randomized, placebo-controlled, double-blind study. Food Chem Toxicol. 2011 Sep;49(9):2356-64. doi: 10.1016/j.fct.2011.06.038. Epub 2011 Jun 21. PMID 21722694
- [Background] Laws GA, Harold LK, Tagg JR, Hale JDF. Interferon Gamma Response in Human Saliva Following Exposure to the Oral Probiotic Streptococcus salivarius BLIS K12. Probiotics Antimicrob Proteins. 2024 Feb;16(1):93-98. doi: 10.1007/s12602-022-10010-0. Epub 2022 Dec 8. PMID 36477439